CLINICAL TRIAL: NCT04484480
Title: Balance and Motion Coordination Parameters Can be Improved in Patients - Non-randomized Controlled Trial
Brief Title: Balance and Motion Coordination Parameters Can be Improved in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Gait DM
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2; Gait Disorders, Neurologic
Keywords: diabetes; gait; balance; falls
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Gait Disorders, Neurologic; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator an outcomes assessor were blinded for the information whether analyzed participant was in the interventional group or control one.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training (Experimental): Patients included in the study group, who received 3-month proprioception, balance and motor coordination training using the dynamic platform - Biodex Balance System.
  Interventions: Procedure: Balance training
- Control group (No Intervention): Patients included in the control group who did not received any intervention

INTERVENTIONS:
Procedure: Balance training — Proprioception, balance and motor coordination training using the dynamic platform - Biodex Balance System.
  Arms: Balance training

SUMMARY:
Diabetes mellitus type II (DMII) causes many complications, including retinopathy and peripheral neuropathy. These complications are well understood and believed to contribute to gait instability and increase the risk of falls. Poor balance control and increased falling risk have also been reported in people with diabetic peripheral neuropathy (DPN).

Patients with DPN are at an increased risk of falling due to the decreased proprioceptive feedbacks. Effective balance training should improve instabilities of postural control in patients with DPN. For this purpose, evaluations and balance training was designed.

The goal of our study was to establish values for proprioception, balance, muscle coordination and strength in patients with DMII, who underwent biofeedback balance training using the Biodex Balance System.

DETAILED DESCRIPTION:
It is estimated that by the end of 2017 year, there will be 462 millions of patients suffering from diabetes mellitus type II (DMII), what is about 6% of world population (4,4% between 15 and 49 years of age, 15% between 50 and 69 years and 22% of patients older than 70 years). It is predicted that by the beginning of 2030, number of cases on 100000 people will grow from 6059 up to 7079. There are studies proving that cardiovascular complications related to the diabetes are responsible for 4 millions of deaths annually. The newest epidemiological data suggest that growing number of DMII cases is no longer a problem in developed countries but also affects developing ones. As potential risk factors, well proved in the literature authors reported alcoholism, nicotinism, high body-mass index (BMI) and positive family history. It is therefore anticipated that the prevalence of one of its common complications, a diabetic peripheral neuropathy (DPN), will increase as well. It is broadly recognized that a DPN leads to a decrement in distal lower limb sensory function; however, there is also a neuropathy-related decrease in distal motor function, even among those with relatively mild diabetic disease. It is well proven in the literature, that diabetes mellitus influences negatively function of peripheral nervous system by damaging sensory fibers. A high risk of falls has been reported in the diabetic population, with an overall incidence of 1.25 falls/person-year.It was proven that short-period strength and balance exercises do not improves diabetic patients quality of life However they have positive influence on the functional outcome of those people. Influence of DMII on motion system is not limited only to the peripheral nervous system. It also affects structures of cerebrum such as: cerebral cortex, cerebellum or basal nuclei. DMII affects motor and somatosensory cerebral atrophy what leads to changes in projection tracts associated with them. In cerebellum it affects on the vermis and parts of lobes responsible for receiving impulses from the spinal cord and controlling proximal parts of muscles, which are crucial for movement coordination during gait. Disorders caused by DMII in basal nuclei result in longer response time and slower gait velocity. Together with pharmacological and dietary interventions, exercise interventions including resistance training, represent the cornerstones of type 2 diabetes management. In addition to the beneficial effects of exercise interventions on glycemic control and on the cardiovascular risk factors associated with type 2 diabetes, physical exercise is an effective intervention to improve muscle strength, power output, cardiovascular function and functional capacity in elderly diabetic patients. In elderly diabetics with severe functional decline, multicomponent exercise programs composed of resistance, endurance, balance and gait retraining should be employed to increase functional capacity and quality of life and to avoid disability and falls. The aim of the study was to evaluate balance and motor coordination parameters in patients treated for type 2 diabetes who received biofeedback-equivalent training using the Biodex dynamometric platform.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* age over 65
* diagnosed type 2 diabetes, subjected to pharmacological treatment (study group)
* no type 2 diabetes (control group)

Exclusion Criteria:

* unwillingness to participate in the study
* age below 65 years
* surgical intervention in the lower limbs or spine during the last 6 months
* symptoms of osteoarthritis or pain of another origin around the lower limbs or spine
* rheumatic diseases (eg. rheumatoid arthritis, ankylosing spondylitis)
* diagnosed neuromuscular disease
* strongly manifested imbalances due to impairment of central or peripheral nervous system
* neurological disorders with dizziness, nystagmus, dermatologic or profound (cerebrospinal syndrome, dizziness, multiple sclerosis, Parkinson's disease, etc.).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Fall risk test | 3-months after inclusion to the study
  Test performed with use of Biodex platform to measure participant's ability to maintain the center of gravity on an unstable substrate in three 20-second trials. The lower the values of the fall index were, the better the result.
General Stability Index | 3-months after inclusion to the study
  Test performed with use of Biodex platform to measure participant's ability to maintain the center of gravity on an unstable substrate in three 20-second trials
Frontal-Posterior Stability Index) | 3-months after inclusion to the study
  Test performed with use of Biodex platform to measure participant's ability to maintain the center of gravity on an unstable substrate in three 20-second trials
Medial-Lateral Stability Index | 3-months after inclusion to the study
  Test performed with use of Biodex platform to measure participant's ability to maintain the center of gravity on an unstable substrate in three 20-second trials

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used during the current study are not publicly available because of patient integrity but are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available on reasonable request for 36 months

REFERENCES:
- [Derived] Adamska O, Mamcarz A, Lapinski M, Radzimowski K, Stepinski P, Szymczak J, Swiercz M, Zarnovsky K, Maciag BM, Stolarczyk A. Continuous glycemia monitoring in perioperative period in patients undergoing total knee or hip arthroplasty: A protocol for a prospective observational study. Medicine (Baltimore). 2022 Oct 21;101(42):e31107. doi: 10.1097/MD.0000000000031193. PMID 36281192
- [Derived] Stolarczyk A, Jarzemski I, Maciag BM, Radzimowski K, Swiercz M, Stolarczyk M. Balance and motion coordination parameters can be improved in patients with type 2 diabetes with physical balance training: non-randomized controlled trial. BMC Endocr Disord. 2021 Jul 3;21(1):143. doi: 10.1186/s12902-021-00804-8. PMID 34217288